CLINICAL TRIAL: NCT04393337
Title: Gestational Age Versus Nasal-tragus Length for Estimating Endotracheal Tube Insertion Depth in Newborns - A Randomised Trial
Brief Title: Estimating Length of Endotracheal Tube Insertion Using Gestational Age or Nasal-Tragus Length in Newborn Infants
Acronym: ELEGANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: King Fahad Hospital (Unknown); King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Abdul Razak, Clinical Assistant Professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-0148
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Endotracheal Tube Tip Position; Bronchopulmonary Dysplasia; Pneumothorax; Death; Duration, Ventilator
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Pneumothorax; Death

STUDY DESIGN:
Intervention Model Description: Eligible infants will be randomly assigned (1:1) to the 'gestational age chart' or 'nasal-tragus length' method We will stratify the randomization by gestational age at birth (<28 weeks and >28 weeks) and participating center. An independent researcher will generate the randomization sequence with a computer at the website www.sealedenvelope.com hosted by King Abdullah bin Abdulaziz University Hospital, Saudi Arabia. The researcher will upload the sequence to the in-built randomization module within the Research Electronic Data Capture (REDCap) system. The sequence is inaccessible to the trial investigators. We will conceal the allocation by incorporating the random permuted blocks of size 2 and 4 sequences within the REDCap system.
Who Masked: Outcomes Assessor
Masking Description: Blinding of the clinicians, nurses, and patient caregivers are impractical. However, to minimize the bias, we will neither mention the method used to estimate the endotracheal tube insertion depth to the patient caregivers explicitly and nor record in the patient charts. We will blind the primary outcome assessment by masking the consultant pediatric radiologist to the group assignment. Similarly, the consultant pediatric radiologist will determine the following secondary outcomes-endotracheal tube tip above the upper border of T1 vertebra, endotracheal tube tip below the lower border of T2 vertebra, and pneumothorax. The other secondary outcomes (endotracheal tube repositioning after the X-ray, oxygen therapy at 28 days, oxygen therapy, or positive pressure support at 36 weeks post-menstrual age, duration of invasive ventilation, and death before discharge) will be determined by the trained research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gestational Age Chart Method (Experimental): In this method, the endotracheal tube insertion depth is obtained from the gestational age chart provided in the 7th edition textbook of neonatal resuscitation program (adapted from Kempley et al. PubMed identifier number: 18372092)
  Interventions: Other: Gestational Age Chart Method
- Nasal-Tragus Length Method (Active Comparator): In this method, the endotracheal tube insertion depth is calculated based on the formula-the distance from nasal septum tip to ear tragus+1 cm
  Interventions: Other: Nasal-Tragus Length Method

INTERVENTIONS:
Other: Gestational Age Chart Method — The endotracheal tube insertion depth is obtained by the gestational age chart
  Arms: Gestational Age Chart Method
Other: Nasal-Tragus Length Method — The endotracheal tube insertion depth is obtained by the nasal-tragus method formula
  Arms: Nasal-Tragus Length Method

SUMMARY:
Endotracheal intubation is a life-saving intervention that few infants need after birth. Although an endotracheal tube is the most reliable way of providing positive-pressure breath, the critical factor that determines the maximal efficacy of positive-pressure ventilation is the optimal placement of the endotracheal tube tip. There are various methods available to determine the initial depth of endotracheal tube (ETT) that are based on the infant's birth weight, gestational age, anthropometric measurements, and others include vocal cord guide and suprasternal palpation methods.

The Neonatal Resuscitation Program (NRP) textbook, in its 7th edition of the textbook, recommends a gestational age chart and nasal-tragus length method for estimating endotracheal tube insertion depth during cardiopulmonary resuscitation of the neonate. The evidence to support these two methods is, however, limited. Hence, we designed this study to determine the accuracy of two methods, gestational age chart and nasal-tragus length method, recommended by the Neonatal Resuscitation Program.

DETAILED DESCRIPTION:
Trial Objective: To determine whether estimating ETT insertion depth using gestational age chart rather than nasal-tragus length method results in more correctly positioned ETT tips.

Setting: The neonates will be recruited from multiple tertiary-level neonatal intensive care units in Saudi Arabia. A neonate can participate in more than one clinical trial, depending on the interventions being given. Parallel run trials will be discussed between the chief and local principal investigators whether or not joint recruitment is feasible to both parties.

Informed Consent: We will obtain written consent after the parents have been given a full verbal explanation and written description. We will explain to the parents in their own native language. We will use a hospital-based adult interpreter wherein required. We will obtain deferred consent (after initial verbal assent) where prior consent is not feasible as the study does not involve additional risk or investigations to the participants, and the interventions are otherwise considered as standard practice recommendations by the NRP.

Data Safety Monitoring Board: Any unexpected serious events (death, any life-threatening event, any event that will prolong the hospitalization or any event that will result in disability) will be reported to the data safety monitoring committee. The trial steering committee will receive recommendations from the data safety monitoring board if the trial requires early termination following the interim data analyses and evidence from relevant studies. The following measures were agreed to consider stopping the trial, wholly or partly (subgroups), after an interim analysis, that will be done after recruiting 200 participants.

1. An absolute difference of greater than or equal to 25% in the primary outcome between the study groups.
2. An absolute difference of less than 5% in the primary outcome between the study groups.
3. A rate of less than 20% in the primary outcome in either of the groups.

Sample Size: Our unpublished data showed using the nasal-tragus length method results in 35% of correctly positioned ETT tips in term and preterm infants. The data is similar to the randomized and non-randomized studies that showed an accuracy between 32 and 37 percent using the nasal-tragus length method. With 90% power and two-sided 5% significance, to detect an absolute increase in optimally positioned ETT tips of 15%, we will require 454 participants. We calculated sample size using nQuery Advisor Sample Size Calculator version 8.3.0.0.

Statistical Analysis: We will analyze the data based on the intention-to-treat principle. Univariate analyses will be performed to compare baseline demographic factors between the two groups. A mean with standard deviation (normal data) or median with interquartile range (skewed data) will be obtained for continuous variables and numbers and percentages for categorical variables. Independent T-test (normal data) or Mann Whitney U test (skewed data) for continuous variables and chi-square test (or Fisher's exact test as appropriate) for categorical variables will be used for analyses between the groups. Statistical Analysis Software version 9.4 will be used for the conduct of all analyses.

Analysis of primary outcome: Adjusted risk ratios of a successful outcome will be calculated along with 95% confidence intervals. Adjusted ratios will be determined by way of multivariable logistic regression analysis, including co-variates deemed biologically to have an influence on the primary outcome (gestational age, small for gestational age, and center). Principles of best model practices will be followed (including assessment of collinearity amongst included variables) as well as the determination of the predictive ability of the model using area under the curve.

Analysis of secondary outcomes: Similar analyses as above will be performed for all secondary outcomes that are categorical variables. The risk ratios of secondary outcomes mortality, oxygen therapy at 28 days, pneumothorax, and bronchopulmonary dysplasia will be adjusted based on the following variables: gestational age, male sex, small for gestational age, maternal hypertension, chorioamnionitis, antenatal steroids, and center if the P-value is less than 0.25 on univariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Infants (less than 28 days of life) between 23 weeks 0 days and 41 weeks 6 days gestational age
* Infants requiring oral intubation in the delivery room or in neonatal intensive care unit

Exclusion Criteria:

* Infants with major chromosomal anomalies, including trisomy 13, trisomy 18, and trisomy 21
* Infants with major anomalies, including craniofacial anomalies and facial dysmorphism that may affect the nasal-tragus length

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 454 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of infants with optimally positioned endotracheal tube tip on the chest X-ray | within 4 hours of endotracheal intubation
  Endotracheal tube tip is considered optimally positioned if the tip lies between upper border of first thoracic vertebra (T1) and the lower border of second thoracic vertebra (T2) on the chest X-ray. While obtaining the antero-posterior view chest X-ray in supine position, the infant's head, neck and chest is placed in the midline with no tension on the endotracheal tube and neck being in neutral position (i.e. neck neither flexed nor extended). Just before obtaining the film, the investigator/research assistant should re-confirm that the endotracheal tube is secured in a standardize manner at the estimated depth based on the treatment arm assigned.

SECONDARY OUTCOMES:
Proportion of infants with endotracheal tube tip above T1 vertebra | within 4 hours of endotracheal intubation
  Presence of endotracheal tube tip above the upper border of first thoracic vertebra e of endotracheal tube tip below the lower border of second thoracic vertebra on the chest X-ray
Proportion of infants with endotracheal tube tip below T2 vertebra | within 4 hours of endotracheal intubation
  Presence of endotracheal tube tip below the lower border of second thoracic vertebra on the chest X-ray
Proportion of infants with pneumothorax | 36 weeks of post-menstrual age
  Presence of air in the pleural space determined by a chest X-ray
Proportion of infants with requiring endotracheal tube repositioning (advance or withdrawn) following chest X-ray | 24 hours
  Repositioning of the endotracheal tube will be done based on attendings discretion
Proportion of infants with oxygen therapy | 28 days from the birth
  Any supplemental oxygen (>21%) on invasive or non-invasive respiratory support
Proportion of infants with bronchopulmonary dysplasia | 36 weeks of post-menstrual age
  It is defined as oxygen therapy or positive pressure support (include nasal cannula <2 liter/minute and >30% oxygen, nasal cannula >2 liters/minute and any oxygen, continuous positive airway pressure and any oxygen, or invasive respiratory support and any oxygen)
Ventilation days | 36 weeks of post-menstrual age
  Duration of invasive ventilation
Proportion of infants with mortality | 36 weeks of post-menstrual age
  Death occurring anytime from birth until discharge

CONTACTS AND LOCATIONS:
Locations (3):
- Saudi Arabia (3):
  - King Fahad Hospital, AlBaha University, Al Bahah
  - King Abdullah bin Abdulaziz University Hospital, Riyadh
  - King Faisal Specialist Hospital & Research Centre, Riyadh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Razak A, Faden M, Alghamdi J, Binmanee A, Alonazi AH, Hamdoun A, Almugaiteeb S, Patel W, Katar H, Lora F, Alismail A, Lavery A, Hamama I, Alsaleem N, Alshaikh M, Alrasheed L, Aldibasi O. Randomised trial estimating length of endotracheal tube insertion using gestational age or nasal-tragus length in newborns: a study protocol. BMJ Open. 2022 Jan 19;12(1):e055628. doi: 10.1136/bmjopen-2021-055628. PMID 35046004